CLINICAL TRIAL: NCT07110389
Title: Effectiveness of a Mobile Application-Based Tele-cardiac Rehabilitation (Tele-CR) Program for Patients With Coronary Heart Disease (CHD): A Randomized Clinical Trial
Brief Title: Effectiveness of a Tele-cardiac Rehabilitation (Tele-CR) Program
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung University of Science and Technology (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government); Chang Gung University (Other); Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 202301928B0-1
Record Dates: First submitted 2025-07-25; First posted 2025-08-07 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Coronary Heart Disease (CHD); Coronary Arterial Disease (CAD)
Keywords: coronary heart disease; cardiac rehabilitation; telemedicine; mobile health
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The tele-cardiac rehabilitation (tele-CR) program for the intervention group and the attention control for the control group were delivered by the same two researchers. Both researchers are clinical specialists with over 20 years of experience in cardiology. One researcher provided the intervention during hospitalization, while the other managed the post-discharge follow-up and mobile application support. Standard care was provided to both groups throughout the study. Data collection was performed by a single research assistant who was blinded to group allocation. Additionally, ward and outpatient clinical staff involved in patient care and outcome data collection were also blinded to participant group assignments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A tele-CR program (Experimental): The six-month tele-cardiac rehabilitation (tele-CR) program consists of three components: motivational interviewing, mobile application (App) implementation, and self-management with follow-up tracking.
  Interventions: Behavioral: A tele-CR program
- Attention-controlled (Other): The control group received regular contact via LINE or telephone for six months following discharge, matched in frequency and duration to the follow-up provided in the intervention group.
  Interventions: Other: Attention-controlled

INTERVENTIONS:
Behavioral: A tele-CR program — The tele-CR program is divided into three parts: motivational interviewing, app delivery, and self-management and tracking. Motivational interviewing was conducted during hospitalization and involved evaluating individual risk factors, setting behavioral goals, and providing training on the installation and operation of the tele-CR app (approximately 30-60 minutes per session).
  After discharge, researchers monitored app usage and conducted seven follow-up sessions via LINE or telephone at 1 week, and at 1, 2, 3, 4, 5, and 6 months post-discharge. These follow-ups, each lasting approximately 5-15 minutes, aimed to assess patients' living conditions, address any issues promptly, and provide encouragement or praise based on their engagement with the app.
  After the completion of the 6-month tele-CR intervention, participants could still actively contact the researchers via LINE or the app to seek health-related assistance according to their personal needs, up to 12 months post-discharge.
  Arms: A tele-CR program
Other: Attention-controlled — The researchers conducted face-to-face communication with participants in the control group prior to discharge, aiming to establish a professional relationship and advise them to follow routine health education and adopt an appropriate lifestyle. After discharge, follow-up care was provided regularly via LINE or telephone at 1 week, and at 1, 2, 3, 4, 5, and 6 months post-discharge-a total of seven sessions, each lasting approximately 3-5 minutes-to inquire about any symptoms of discomfort.
  Arms: Attention-controlled

SUMMARY:
This study represents the second phase of a three-year research project aimed at evaluating both the short- and long-term effects of a six-month tele-cardiac rehabilitation (tele-CR) program in patients with coronary heart disease (CHD). The primary outcomes include quality of life, self-efficacy, self-management, medication adherence, and mental health (anxiety and depression). In addition, comprehensive metabolic parameters will be assessed, including body mass index (BMI), systolic and diastolic blood pressure (SBP and DBP), fasting blood glucose (FBG), glycosylated hemoglobin (HbA1C), and lipid profile markers such as triglycerides (TG), total cholesterol (TC), high-density lipoprotein (HDL), and low-density lipoprotein (LDL).

DETAILED DESCRIPTION:
Coronary heart disease (CHD) is a leading cause of death in Taiwan and a major contributor to premature and avoidable mortality worldwide. Cardiac rehabilitation (CR) is a multidisciplinary secondary prevention strategy that has been widely proven to reduce morbidity and mortality. However, despite its well-documented benefits, CR remains underutilized due to barriers such as transportation, time constraints, and limited access to facilities. Tele-cardiac rehabilitation (tele-CR), a technology-enabled alternative to traditional center-based CR, has been shown to be both safe and effective in improving clinical and behavioral outcomes. Nevertheless, research on the implementation and effectiveness of tele-CR in Taiwan is still limited.

This project spans a three-year period and is divided into two phases. The present study represents the second phase and aims to evaluate the short- and long-term effects of a six-month tele-CR program in patients with CHD. The primary outcomes include quality of life, self-efficacy, self-management, medication adherence, and mental health status (anxiety and depression). In addition, a comprehensive set of metabolic parameters will be assessed, including BMI, SBP, DBP, FBG, HbA1C, and lipid profile markers such as TG, TC, HDL, and LDL.

The research hypotheses are as follows: the tele-CR program will (1) improve quality of life, self-efficacy, self-management, and medication adherence; (2) reduce levels of anxiety and depression; and (3) lower blood pressure, blood glucose, BMI, and lipid levels, with these effects being sustained up to 12 months post-discharge.

A single-blind, attention-controlled, prospective, randomized clinical trial will be conducted in the cardiology ward of a medical center in northern Taiwan from September 1, 2025, to August 31, 2027. A total of 126 patients diagnosed with CHD will be purposively recruited upon admission. After completing baseline assessments, participants will be randomly assigned in blocks to either the experimental group (n = 63) or the control group (n = 63). The experimental group will participate in a six-month tele-CR program, consisting of in-hospital motivational interviews, mobile application support, self-management education, and seven scheduled follow-up calls. The control group will receive standard care plus seven routine care calls over the same six-month period following discharge. Both groups will continue to receive usual medical and nursing care throughout the study.

This study has been reviewed and approved by the Institutional Review Board (IRB) of the study hospital. Research assistants will explain the study's objectives and procedures in detail to all eligible participants. Informed written consent will be obtained only after participants' questions have been addressed. Questionnaire data will be collected either via self-administration or with assistance from trained research personnel, based on participant preference. All data collection will take place in a quiet and private environment to ensure accuracy and participant comfort.

Data will be collected at baseline and at 3, 6, 9, and 12 months after discharge, using structured questionnaires and medical records. Baseline values for metabolic indicators will be based on the closest hospitalization date within the three months prior to admission. Post-discharge values will be based on the closest record to the date of each questionnaire completion.

All statistical analyses will be performed using SPSS version 26.0. Descriptive statistics (frequencies, percentages, means, and standard deviations) will summarize the participant characteristics and study variables. An intention-to-treat approach will be adopted. To examine the short- and long-term effects of the intervention, generalized estimating equations (GEE) will be used. A two-tailed test with a significance level of p < 0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

1. The main diagnosis at admission of CHD.
2. Age ≥20 years.
3. Owns an iOS or Android smartphone and can use it.
4. Conscious, clear and can communicate.
5. Agrees to participate in the research after explanation and is willing to use the App.

Exclusion Criteria:

1. Level IV on the New York Heart Association Functional Classification.
2. Left ventricular ejection fraction<40%.
3. Have a history of severe arrhythmia (e.g., ventricular tachycardia, ventricular fibrillation, complete atrioventricular block).
4. Combined with other serious heart diseases (e.g., congenital heart disease, cardiomyopathy).
5. Mental disorders, end-stage renal disease and other systemic diseases diagnosed by a physician.
6. Severe infection, injury, surgery (e.g., coronary artery bypass graft) or cancer treatment has occurred in the past three months.
7. Physical activities are affected by neurological, respiratory, skeletal, or peripheral vascular diseases.
8. Restricted use of the App due to sensory or cognitive impairment.
9. Already participated in other clinical trials.
10. Planning to receive surgery (e.g., coronary artery bypass graft).

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Level of health-related quality of life | baseline, and 3, 6, 9, 12 months after discharge
  The Chinese version of the Seattle Angina Questionnaire (SAQ), translated by Tsai and Chie (2002), is used to assess participants' health-related quality of life over the past month. The questionnaire consists of 19 items covering five domains. Each question is scored using an ordinal scale, and each aspect is converted into [(total score of the aspect question - minimum total score)/scoring range * 100] from 0 to 100 points, with higher scores indicating better status in that domain. In this study, the average of three domains-physical activity, angina frequency, and disease perception (each with a score range of 0-100)-is considered the overall SAQ score. A higher total score reflects better overall health-related quality of life (Patel et al., 2018). The test-retest reliability of the Chinese version of the SAQ over 3 to 4 weeks ranges from 0.44 to 0.79; internal consistency ranges from 0.43 to 0.84; and criterion-related validity ranges from 0.44 to 0.84 (Tsai and Chie, 2002).
Level of general quality of life | baseline, and 3, 6, 9, 12 months after discharge
  The EuroQol-5-Dimensions-5-Level (EQ-5D-5L) is a widely used generic quality-of-life scale that has been translated into multiple languages and has demonstrated good reliability and validity (EuroQol Research Foundation, 2019; Feng et al., 2021). The five-digit health state profiles are converted into a utility value using a set of weights derived from a Taiwanese population study, ensuring suitability for the Chinese population. The utility value ranges from -1.0259 to 1, where lower values indicate poorer health-related quality of life (Lin et al., 2018). The second component of the EQ-5D-5L is a visual analog scale (VAS) ranging from 0 to 100, where higher scores reflect better self-perceived quality of life (EuroQol Research Foundation, 2019).

SECONDARY OUTCOMES:
Level of self-efficacy and self-management | baseline, and 3, 6, 9, 12 months after discharge
  This study used the Chinese version of the Heart Health Self-Efficacy and Self-Management (HH-SESM) scale, translated and revised by Wu et al. (2022). The scale comprises 12 items covering domains such as physical activity, diet, medication, psychosocial factors, weight management, and smoking. Each item includes two parts: self-efficacy and self-management. The self-efficacy subscale asks, "How confident are you that you can do the following?", while the self-management subscale asks, "How often do you do the following?" Both are scored using a 4-point Likert scale. Higher total scores indicate greater levels of self-efficacy and self-management. The internal consistency of the Chinese version of the HH-SESM ranges from 0.72 to 0.77; the two-week test-retest reliability ranges from 0.71 to 0.76; the split-half reliability is between 0.79 and 0.80; and the explained variance ranges from 25.2% to 31.1% (Wu et al., 2022).
Level of medication adherence | baseline, and 3, 6, 9, 12 months after discharge
  The 8-item version Morisky Medication Adherence Scale (MMAS-8) consists of 8 items. Each of the first 7 items has 2 possible responses (yes/no), while the 8th item is answered with a 5-point Likert scale. The possible total medication adherence score ranges between 0 and 8, and the higher the score, the better the adherence level. A total score < 6 isconsidered low adherence, while a total score of ≥ 6 but < 8 indicates moderate adherence, and a scoreof 8 indicates high adherence (Berlowitz et al., 2017; Bress et al., 2017). The original MMAS-8 has demonstrated good reliability and validity (Moon et al., 2017). For the Chinese version, internal consistency ranges from 0.65 to 0.83, explaining approximately 46% of the variance, with a test-retest correlation coefficient of 0.80 (Ho & Lee, 2014; Wang et al., 2013).
Level of anxiety and depression | baseline, and 3, 6, 9, 12 months after discharge
  The original version of the Hospital Anxiety and Depression Scale (HADS) was developed by Zigmond and Snaith in 1983. The Chinese version of the HADS is used to assess anxiety and depression symptoms experienced by individuals over the past week. It consists of 14 items, with 7 items measuring anxiety and 7 items measuring depression. Each item is rated on a four-point scale (0-3), yielding subscale scores ranging from 0 to 21. Higher scores indicate more severe levels of anxiety or depression. The internal consistency of the Chinese version of the HADS ranges from 0.77 to 0.82, and the one-week test-retest reliability ranges from 0.64 to 0.83 (Chen et al., 1999).
Body Mass Index (BMI) | baseline, and 3, 6, 9, 12 months after discharge
  Values will be extracted from medical records. The baseline value will be based on the closest hospitalization date within the three months before hospitalization. The post-discharge value will be based on the closest questionnaire filling date (i.e., at 3, 6, 9, and 12 months after discharge). BMI will be calculated using body weight (in kilograms) and height (in meters) according to the formula: BMI = weight (kg) / [height (m)]².
  Unit of measure: Kilograms per square meter (kg/m²).
Systolic Blood Pressure (SBP) | baseline, and 3, 6, 9, 12 months after discharge
  Values will be extracted from medical records. The baseline value will be based on the closest hospitalization date within the three months before hospitalization. The post-discharge value will be based on the closest questionnaire filling date (i.e., at 3, 6, 9, and 12 months after discharge).
  Unit of measure: Millimeters of mercury (mmHg).
Diastolic Blood Pressure (DBP) | baseline, and 3, 6, 9, 12 months after discharge
  Values will be extracted from medical records. The baseline value will be based on the closest hospitalization date within the three months before hospitalization. The post-discharge value will be based on the closest questionnaire filling date (i.e., at 3, 6, 9, and 12 months after discharge).
  Unit of measure: Millimeters of mercury (mmHg).
Fasting Blood Glucose (FBG) | baseline, and 3, 6, 9, 12 months after discharge
  Values will be extracted from medical records. The baseline value will be based on the closest hospitalization date within the three months before hospitalization. The post-discharge value will be based on the closest questionnaire filling date (i.e., at 3, 6, 9, and 12 months after discharge).
  Unit of measure: Milligrams per deciliter (mg/dL).
Glycosylated Hemoglobin (HbA1c) | baseline, and 3, 6, 9, 12 months after discharge
  Values will be extracted from medical records. The baseline value will be based on the closest hospitalization date within the three months before hospitalization. The post-discharge value will be based on the closest questionnaire filling date (i.e., at 3, 6, 9, and 12 months after discharge).
  Unit of measure: Percentage (%).
Triglycerides (TG) | baseline, and 3, 6, 9, 12 months after discharge
  Values will be extracted from medical records. The baseline value will be based on the closest hospitalization date within the three months before hospitalization. The post-discharge value will be based on the closest questionnaire filling date (i.e., at 3, 6, 9, and 12 months after discharge).
  Unit of measure: Milligrams per deciliter (mg/dL).
Total Cholesterol (TC) | baseline, and 3, 6, 9, 12 months after discharge
  Values will be extracted from medical records. The baseline value will be based on the closest hospitalization date within the three months before hospitalization. The post-discharge value will be based on the closest questionnaire filling date (i.e., at 3, 6, 9, and 12 months after discharge).
  Unit of measure: Milligrams per deciliter (mg/dL).
High-Density Lipoprotein (HDL) | baseline, and 3, 6, 9, 12 months after discharge
  Values will be extracted from medical records. The baseline value will be based on the closest hospitalization date within the three months before hospitalization. The post-discharge value will be based on the closest questionnaire filling date (i.e., at 3, 6, 9, and 12 months after discharge).
  Unit of measure: Milligrams per deciliter (mg/dL).
Low-Density Lipoprotein (LDL) | baseline, and 3, 6, 9, 12 months after discharge
  Values will be extracted from medical records. The baseline value will be based on the closest hospitalization date within the three months before hospitalization. The post-discharge value will be based on the closest questionnaire filling date (i.e., at 3, 6, 9, and 12 months after discharge).
  Unit of measure: Milligrams per deciliter (mg/dL).

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung University of Science and Technology, Taoyuan District, Guishan Dist., Taiwan

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because the study involves sensitive health information, and the informed consent obtained from participants does not include permission for public sharing of individual-level data. Data sharing is also restricted by applicable privacy laws and institutional policies to protect participant confidentiality.